CLINICAL TRIAL: NCT01449955
Title: mTOR Kinase as a Therapeutic Target in Reconsolidation of Posttraumatic Stress Disorder-related Traumatic Memory
Brief Title: Rapamycin as a Means of Interference With Reconsolidation of Posttraumatic Stress Disorder-related Traumatic Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alina Suris, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-049
Record Dates: First submitted 2011-09-16; First posted 2011-10-10 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sirolimus; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (e.g., sugar pill) (Placebo Comparator): 15 mg Placebo will be administered once, in pill form.
  Interventions: Drug: Placebo
- Rapamycin (Active Comparator): 15 mg of Rapamycin will be administered once, in pill form.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Sirolimus is an FDA approved immunosuppressant drug used to prevent rejection in organ transplantation, and is especially useful in kidney transplants. It is non-toxic to kidneys, unlike other immunosuppressants. In this study, the medication will be administered once to see if it interferes with emotional memory reconsolidation. This is based on the fact that it inhibits the mammalian target of Rapamycin (mTOR) through directly binding the mTOR Complex1 (mTORC1). mTOR is a serine/threonine protein kinase that regulates cell growth, cell proliferation, cell motility, cell survival, protein synthesis and transcription.
  a single dosage of 15mg will be administered during this study.
  Other Names: Sirolimus; X-Rapamune
  Arms: Rapamycin
Drug: Placebo — Inactive
  Other Names: sugar pill
  Arms: Placebo (e.g., sugar pill)

SUMMARY:
The purpose of the proposed study is to determine if pairing reactivation of a traumatic memory with a single administration of Rapamycin (e.g., Sirolimus) in men with combat-related Posttraumatic Stress Disorder leads to a reduction of the emotional strength of that particular traumatic memory.

The following hypotheses will be tested:

1. Traumatic memory reactivation paired with a single dose of Rapamycin will decrease objective measures of stress and self-report of stress during replay of the traumatic memory, relative to, subjects receiving placebo.
2. Pairing administration of Rapamycin with traumatic memory reactivation will decrease symptoms of Posttraumatic Stress Disorder one month and three months later, relative to patients receiving placebo.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is characterized by intrusive memories in the form of unwanted images, nightmares, and flashbacks as the result of being exposed to a traumatic event . Current research efforts have begun to explore the underlying neurochemical changes associated with PTSD. Recently, these efforts have focused on the prevention of PTSD in persons exposed to trauma. For example, preliminary evidence suggests that interference with consolidation of trauma-related memories using the beta-antagonist, propranolol, may prevent PTSD in humans with recent traumas. However, given that as much as 90% of the US population is exposed to at least one traumatic event during their lifetimes, the utility of this treatment is limited by the logistical problems of treating everyone at risk. To date, there have been very few systematic studies on humans that focus on changing the underlying traumatic memory once PTSD has been established.

The trauma experience is initially stored in short-term memory, then consolidated into long-term memory. However, the long-term stability conferred by the consolidation process undergoes a period of labiality as follows. Each time a consolidated memory is activated, the memory trace becomes newly labile and must be consolidated again to remain in long-term memory5. This process is called reconsolidation. Reconsolidation therefore offers a biologic window during which long-term memories can be disrupted. Preclinical studies have begun to unravel the biological changes that underlie these processes. Both pharmacological agents, including glucocorticoids, and protein synthesis inhibitors can interfere with memory consolidation and reconsolidation. In preclinical studies, the global protein synthesis inhibitor anisomycin can block reconsolidation, leading to a reduction in strength of traumatic memories. Unfortunately, the toxicity of anisomycin is prohibitive for therapeutic use. Thus, rather than using a global protein synthesis inhibitor, a more effective and selective means of reducing consolidation of an established traumatic memory is to target only a subset of protein translation important for synaptic plasticity. The protein kinase mTOR (mammalian target of rapamycin) is just such a regulator of a subset of protein synthesis critical for synaptic plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans
* Diagnosis of Posttraumatic Stress Disorder related to combat

Exclusion Criteria:

* Hypersensitivity to Rapamycin
* Organic brain damage (including unresolved Traumatic Brain Injury sequela)
* Substance dependence in the last three months
* On any immunosuppressant therapy
* Prominent suicidal or homicidal features
* Medical conditions: systemic infections, congestive heart failure, renal failure, hepatic failure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina M Suris, Ph.D., Principal Investigator — UT Southwestern Medical Center; VA North Texas Healthcare System; Carol North, M.D., Study Chair — UT Southwestern Medical Center; VA North Texas Healthcare System
Locations (1):
- VA North Texas Healthcare System, Dallas, Texas, United States

REFERENCES:
- [Background] Blundell J, Kouser M, Powell CM. Systemic inhibition of mammalian target of rapamycin inhibits fear memory reconsolidation. Neurobiol Learn Mem. 2008 Jul;90(1):28-35. doi: 10.1016/j.nlm.2007.12.004. Epub 2008 Mar 7. PMID 18316213
- [Result] Suris A, Smith J, Powell C, North CS. Interfering with the reconsolidation of traumatic memory: sirolimus as a novel agent for treating veterans with posttraumatic stress disorder. Ann Clin Psychiatry. 2013 Feb;25(1):33-40. PMID 23376868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited by flyers, clinician referral and letters mailed to male VA North Texas patients with PTSD.
Pre-assignment Details: excluded if did not meet PTSD criteria according to the CAPS
Groups:
- Rapamycin (e.g., Sirolimus): 15mg Rapamycin administered once in pill form
- Placebo: 15mg Placebo administered once in pill form
Period: Overall Study
Arm/Group | Rapamycin (e.g., Sirolimus) | Placebo
Started | 28 | 26
Completed | 27 | 24
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Male Veterans with PTSD
Groups:
- Rapamycin: 15mg Rapamycin administered once in pill form
- Total: Total of all reporting groups
Arm/Group | Rapamycin | Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.64 (14.39) | 42.15 (15.46) | 42.21 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 26 | 54
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered Posttraumatic Stress Disorder Scale (CAPS)
Description: Clinician administered interview which assesses the symptoms of Posttraumatic Stress disorder at baseline, and then again 1 month posttreatment. The CAPS is a 25 item semi-structured interview that assesses the 17 DSM-IV PTSD criteria as well as social and occupational impairment. For each item the participant can respond with a rating of 0-8 (with 0 indicating no symptom severity and frequency and 8 indicating extreme symptom severity and frequency). The range of total scores on a CAPS is from 0-136, with a greater score indicating greater PTSD symptom severity. The total score is computed by summing the aforementioned 17 items. Additionally, the CAPS assesses for a positive PTSD diagnosis by assessing for the three DSM-IV criteria of B, C, and D. In order to meet a positive screen for each criteria, a person must screen positive for symptoms by reporting a score of 3 or more on the specific symptom criterion.
Time Frame: Baseline and 1 month posttreatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo: 15 mg Placebo administered once in pill form
Arm/Group | Rapamycin (e.g., Sirolimus) | Placebo
Number analyzed (Participants) | 27 | 24
scores on a scale
  Baseline | 72.13 (15.27) | 70.63 (16.37)
  1 month posttreatment | 58.27 (22.96) | 64.54 (17.88)
Statistical Analysis 1: Comparison: Rapamycin (e.g., Sirolimus) vs Placebo; ANOVA comparing the results of change over time (e.g., comparing baseline to 1 month posttreatment) as well as comparing differences between condition (e.g., placebo compared to rapamycin); Test type: Superiority or Other; p > 0.05, ANOVA

2. Primary Outcome: Clinician Administered Posttraumatic Stress Disorder Scale (CAPS)
Description: The CAPS is administered to assess the frequency and intensity of PTSD symptoms at baseline, and then again 3 months posttreatment. The CAPS is a 25 item semi-structured interview that assesses the 17 DSM-IV PTSD criteria as well as social and occupational impairment. For each item the participant can respond with a rating of 0-8 (with 0 indicating no symptom severity and frequency and 8 indicating extreme symptom severity and frequency). The range of total scores on a CAPS is from 0-136, with a greater score indicating greater PTSD symptom severity. The total score is computed by summing the aforementioned 17 items. Additionally, the CAPS assesses for a positive PTSD diagnosis by assessing for the three DSM-IV criteria of B, C, and D. In order to meet a positive screen for each criteria, a person must screen positive for symptoms by reporting a score of 3 or more on the specific symptom criterion.
Time Frame: change in CAPS score from baseline to 3 months posttreatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rapamycin (e.g., Sirolimus) Baseline: 15mg Rapamycin administered once in pill form at baseline
- Placebo at Baseline: 15 mg Placebo administered once in pill form at baseline
- Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment: 15mg Rapamycin administered once in pill form at 3 months Posttreatment
- Placebo at 3 Months Posttreatment: 15 mg Placebo administered once in pill form at 3 months posttreatment
Arm/Group | Rapamycin (e.g., Sirolimus) Baseline | Placebo at Baseline | Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment | Placebo at 3 Months Posttreatment
Number analyzed (Participants) | 27 | 24 | 27 | 24
units on a scale | 72.13 (15.27) | 70.63 (16.37) | 55.26 (22.62) | 62.63 (17.60)
Statistical Analysis 1: Comparison: Rapamycin (e.g., Sirolimus) Baseline vs Placebo at Baseline vs Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment vs Placebo at 3 Months Posttreatment; Test type: Superiority; p > 0.5, ANOVA

3. Secondary Outcome: PTSD Checklist (PCL)
Description: Self-report instrument which assesses the intensity of Posttraumatic Stress Disorder symptoms. The PCL measures the 17 DSM-IV PTSD criteria in 17 items. For each item the participant can respond with a rating of 1-5 (with 1 indicating not at all bothered 5 indicating extremely bothered by the symptom) The range of total scores on the PCL is from 17-85, with a greater score indicating greater PTSD symptom severity. The total score is computed by summing the aforementioned 17 items.
Time Frame: change in PCL score from baseline to 1 month posttreatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rapamycin (e.g., Sirolimus) at 1 Month Posttreatment: 15mg Rapamycin administered once in pill form at 1 month Posttreatment
- Placebo at 1 Month Posttreatment: 15 mg Placebo administered once in pill form at 1 month Posttreatment
Arm/Group | Rapamycin (e.g., Sirolimus) Baseline | Placebo at Baseline | Rapamycin (e.g., Sirolimus) at 1 Month Posttreatment | Placebo at 1 Month Posttreatment
Number analyzed (Participants) | 27 | 24 | 27 | 24
units on a scale | 57.19 (10.61) | 60.83 (10.26) | 49.62 (13.14) | 55.00 (11.85)
Statistical Analysis 1: Comparison: Rapamycin (e.g., Sirolimus) Baseline vs Placebo at Baseline vs Rapamycin (e.g., Sirolimus) at 1 Month Posttreatment vs Placebo at 1 Month Posttreatment; Test type: Superiority; p > .05, ANOVA

4. Secondary Outcome: PTSD Checklist (PCL)
Description: as for outcome 3
Time Frame: change in PCL score from baseline to 3 months posttreatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rapamycin (e.g., Sirolimus) Baseline | Placebo at Baseline | Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment | Placebo at 3 Months Posttreatment
Number analyzed (Participants) | 27 | 24 | 27 | 24
units on a scale | 57.19 (10.61) | 60.83 (10.26) | 51.07 (13.81) | 54.13 (11.23)
Statistical Analysis 1: Comparison: Rapamycin (e.g., Sirolimus) Baseline vs Placebo at Baseline vs Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment vs Placebo at 3 Months Posttreatment; Test type: Superiority; p > .05, ANOVA

5. Secondary Outcome: Quick Inventory of Depressive Symptomatology (QIDS)
Description: The QIDS is a 16-item self-report measure that assesses how much a participant endorses each of the DSM-IV-TR symptoms of depression, with each item scored from 0 (no endorsement of symptom) to 3 (endorsement of severe symptomatology). Scores on the QIDS range from 0-27, with higher scores indicating higher depressive symptom severity.
Time Frame: change in QIDS score from baseline to 1 month posttreatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rapamycin (e.g., Sirolimus) Baseline | Placebo at Baseline | Rapamycin (e.g., Sirolimus) at 1 Month Posttreatment | Placebo at 1 Month Posttreatment
Number analyzed (Participants) | 27 | 24 | 27 | 24
units on a scale | 14.48 (3.97) | 13.79 (4.45) | 11.27 (5.03) | 11.75 (3.75)
Statistical Analysis 1: Comparison: Rapamycin (e.g., Sirolimus) Baseline vs Placebo at Baseline vs Rapamycin (e.g., Sirolimus) at 1 Month Posttreatment vs Placebo at 1 Month Posttreatment; Test type: Superiority; p < .05, ANOVA

6. Secondary Outcome: Quick Inventory of Depressive Symptomatology (QIDS)
Description: as for outcome 5
Time Frame: change in QIDS score from baseline to 3 months posttreatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rapamycin (e.g., Sirolimus) Baseline | Placebo at Baseline | Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment | Placebo at 3 Months Posttreatment
Number analyzed (Participants) | 27 | 24 | 27 | 24
units on a scale | 14.48 (3.97) | 13.79 (4.45) | 11.56 (5.13) | 11.29 (4.32)
Statistical Analysis 1: Comparison: Rapamycin (e.g., Sirolimus) Baseline vs Placebo at Baseline vs Rapamycin (e.g., Sirolimus) at 3 Months Posttreatment vs Placebo at 3 Months Posttreatment; Test type: Superiority; p > .05, ANOVA

ADVERSE EVENTS:
Groups:
- Rapamycin: 15mg Rapamycin
- Placebo: Placebo arm
Arm/Group | Rapamycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26

LIMITATIONS AND CAVEATS:
Timing of medication administration may not have been optimal and relatively small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes